CLINICAL TRIAL: NCT02069444
Title: Comparison of the Effects of Truview Laryngoscopy and Macintosh Larygonscopy on Intubation Difficulty Score, Intubation Duration and Intubation Quality in Pediatric Patients Between 2-12 Years
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, CIGDEM YILDIRIM GUCLU, specialist anesthesiologist, Ankara University
Other Study IDs: 2-12
Record Dates: First submitted 2014-02-20; First posted 2014-02-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: All the Pediatric Patients Needed Intubation for Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Truview EVO2 laryngoscope: patients intubated withTruview EVO2 laryngoscope
  Interventions: Procedure: Truview EVO2 laryngoscope
- Macintosh laryngoscope: patients intubated with Macintosh laryngoscope
  Interventions: Procedure: Macintosh laryngoscope

INTERVENTIONS:
Procedure: Macintosh laryngoscope — intubation criterias withMacintosh laryngoscopein pediatric patients
  Groups: Macintosh laryngoscope
Procedure: Truview EVO2 laryngoscope — intubation criterias with Truview EVO2 laryngoscope in pediatric patients
  Groups: Truview EVO2 laryngoscope

SUMMARY:
For endotracheal entubation in children mostly Miller and Macintosh blades have been used. On the other hand Truview EVO2 laringoscopes can maintain a better laryngeal view without having a direct sight of the airway and without having to align oral, pharyngeal, and tracheal axes. The aim of this study is to compare the Truview EVO2 laryngoscope and Macintosh laryngoscope in terms of intubation difficulty score, time to intubation and intubation quality score.

ELIGIBILITY:
Inclusion Criteria:

* aged 2-12 pediatric patients

Exclusion Criteria:

* any allergy
* difficult airway history

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric patients undergoing surgery which needs intubation
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-01; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
ease laryngoscopy in children | during laryngoscopy

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara University, Ankara
  - Ankara University, Pediatric Surgery, Ankara